CLINICAL TRIAL: NCT00750243
Title: A Double-Blind, Randomized, Active Comparator Study of LT-NS001 Versus Naprosyn for Seven Days in Healthy Subjects With Endoscopic Evaluation
Brief Title: Comparator Study of LT-NS001 in Healthy Subjects With Endoscopic Evaluation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Logical Therapeutics (Industry)
Responsible Party: K. Lea Sewell, M.D., Logical Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: LT-NS001-002
Record Dates: First submitted 2008-09-08; First posted 2008-09-10 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
MeSH Terms: interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: LT-NS001
- B (Active Comparator)
  Interventions: Drug: Naprosyn®

INTERVENTIONS:
Drug: LT-NS001 — 1200 mg b.i.d. p.o. for 7.5 days
  Arms: A
Drug: Naprosyn® — 500 mg b.i.d. p.o. for 7.5 days
  Arms: B

SUMMARY:
The purpose of this study is to compare naproxen plasma levels and gastroduodenal mucosal injury after administration of LT-NS001 as compared to Naprosyn in subjects age 45-70.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30 kg/m2
* No NSAID's for 14 days prior to baseline endoscopy

Exclusion Criteria:

* Pregnant/Nursing women
* History of documented gastroduodenal ulcer

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Assessment of GI mucosal injury by endoscopy | 7 days

SECONDARY OUTCOMES:
Comparison of naproxen PK at steady state | 7.5 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Goldstein JL, Jungwirthova A, David J, Spindel E, Bouchner L, Pesek F, Searle S, Skopek J, Grim J, Ulc I, Sewell KL. Clinical trial: endoscopic evaluation of naproxen etemesil, a naproxen prodrug, vs. naproxen - a proof-of-concept, randomized, double-blind, active-comparator study. Aliment Pharmacol Ther. 2010 Nov;32(9):1091-101. doi: 10.1111/j.1365-2036.2010.04442.x. Epub 2010 Aug 23. PMID 20804454